CLINICAL TRIAL: NCT03556774
Title: Boosting Chinese Healthcare Service Providers' Utilization of Behavioral and Pharmacotherapy Interventions for Cigarette Smoking Cessation by 'WeChat WeQuit' Program
Brief Title: Boosting Chinese Healthcare Service Providers' Utilization of Smoking Cessation Interventions by 'WeChat WeQuit' Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Yanhui Liao, Attending Psychiatrist, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017S094
Record Dates: First submitted 2018-04-29; First posted 2018-06-14 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation Intervention; Smoking Abstinence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With smoking cessation training (Experimental): Participants who allocate to the intervention group will receive regular smoking cessation training program messages by professional team. One to six messages will be sent per day for 8 weeks. Hand copy of behavioral and pharmacotherapy interventions manual will send to each HSP by mail after randomization. One to three messages will be sent per week until the end of the 1-year follow-up. They will also be encouraged to communicate the experience of using behavioral and pharmacotherapy interventions in their group.
  Interventions: Behavioral: 'WeChat WeQuit' smoking cessation training program
- Without smoking cessation training (No Intervention): Control group participants will not receive any smoking cessation messages by professional team. They will receive messages of thanking them for being in the study and reminding them of the time until 52-week follow-up. One to six messages will be sent per week for 8 weeks. They will be encouraged to communicate the experience of helping patients quit smoking in their group.

INTERVENTIONS:
Behavioral: 'WeChat WeQuit' smoking cessation training program — Providing 'WeChat WeQuit' smoking cessation training program for healthcare service providers (HSPs) and assessing their utilization of behavioral and pharmacotherapy interventions for cigarette smoking cessation.
  Arms: With smoking cessation training

SUMMARY:
In this single-blind, randomized trial, undertaken in China with 8-week interventions and follow-up to 52 weeks, about 2,200 providers will be randomly allocated to the intervention or control group.

DETAILED DESCRIPTION:
Previous studies have been showed that providing behavioral and pharmacotherapy interventions for cigarette smoking patients was effective but rare among Chinese healthcare service providers. In order to minimize the huge gap between the shortage and demand for smoking cessation training program and smoking cessation service, this 'WeChat WeQuit' smoking cessation training program has been designed to assess whether it will increase Chinese healthcare service providers' utilization of behavioral and pharmacotherapy interventions for cigarette smoking cessation or not.

In this single-blind, randomized trial, about 2200 HSPs will be randomly selected (by randomizeR, https://CRAN.R-project.org/package=randomizeR) to 8-week intervention (behavioral and pharmacotherapy interventions for cigarette smoking patients to help them quit smoking) group or control group that only communicates without any standard smoking cessation practices related messages, and follow-up to 52 weeks. The trial will be carried out in into two phases, the first phase is the pilot study (n=200, 8-week intervention and follow-up to 16 weeks) and the second is the main study (n=2000, 8-week intervention and follow-up to 52 weeks). It is hypothesized that 'WeChat WeQuit' training program will improve Chinese HSPs' utilization of behavioral and pharmacotherapy interventions for cigarette smoking cessation and increase quit rate for smoking patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese-speaking healthcare service providers
2. Know how to use WeChat
3. Use WeChat on a daily basis
4. Willing to provide informed consent to participate in the study -

Exclusion Criteria:

1. Non-Chinese speakers
2. Not healthcare service providers
3. Do not use WeChat
4. Unwilling to participate in the study -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of 'WeChat WeQuit' training program. | 52 weeks
  The utilization rate (i.e. rate=smokers treated divided by smokers seen) of behavioral and pharmacotherapy interventions by HSP for smoking patients from 8 to 52-week.

SECONDARY OUTCOMES:
Prevalence of smoking abstinence | 24 weeks
  The proportion of smoking patients with 7-day point prevalence smoking abstinence (not even a puff of smoke, for the last 7 days) at 4, 8, 12, 16, 20 and continuously abstinence assessed at 24-weeks follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanhui Liao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Peng P, Wu Z, Liu Y, Wang C, Tang J, Liao Y. Boosting Smoking Cessation Intervention Utilization in Chinese Health Care Providers: A Randomized Controlled Trial of the "WeChat WeQuit" Medical Education Program. Nicotine Tob Res. 2024 Dec 23;27(1):61-72. doi: 10.1093/ntr/ntae166. PMID 39083005